CLINICAL TRIAL: NCT03800186
Title: The Influence of Ageing on the Incidence and Site of Trauma Femoral Fractures: a Cross-sectional Analysis
Brief Title: Influence of Age on Trauma Femoral Fractures
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CDRPG8H0011
Record Dates: First submitted 2019-01-06; First posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: FEMORAL FRACTURES
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trauma femoral fracture: Patients to be aged ≥20 years and hospitalized for the treatment of femoral fracture following injury. Patients were grouping into five subgroups as patients with fracture of proximal type A, proximal type B, proximal type C, femoral shaft, and distal femur.
  Interventions: Other: Proximal type A; Other: Proximal type B; Other: Proximal type C; Other: femoral shaft; Other: distal femur

INTERVENTIONS:
Other: Proximal type A — Patients with fracture of proximal type A
Other: Proximal type B — Patients with fracture of proximal type B
Other: Proximal type C — Patients with fracture of proximal type C
Other: femoral shaft — Patients with fracture of femoral shaft
Other: distal femur — Patients with fracture of distal femur

SUMMARY:
This study aimed to determine the influence of ageing on the incidence and site of femoral fractures in trauma patients, by taking the sex, body weight, and trauma mechanisms into account.

DETAILED DESCRIPTION:
This retrospective study reviewed data from adult trauma patients aged ≥ 20 years who were admitted into a Level I trauma center, between January 1, 2009 and December 31, 2016. According to the femoral fracture locations, 3859 adult patients with 4011 fracture sites were grouped into five subgroups: proximal type A (n = 1,359), proximal type B (n= 1,487), proximal type C (n = 59), femoral shaft (n = 640), and distal femur (n = 466) groups. A multivariate logistic regression analysis was applied to identify independent effects of the univariate predictive variables on the occurrence of fracture at a specific site. The propensity score accounts for the risk of a fracture at a specific femoral site was calculated and presented visually with age in a two-dimensional plot.

ELIGIBILITY:
Inclusion Criteria:

* Patients to be aged ≥20 years and hospitalized for the treatment of femoral fracture following injury

Exclusion Criteria:

* Patients with incomplete data were excluded

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study reviewed data from 27,462 trauma patients registered between January 1, 2009 and December 31, 2016. The inclusion criteria required patients to be aged ≥20 years and hospitalized for the treatment of femoral fracture following injury. Patients with incomplete data were excluded.
Sampling Method: Probability Sample
Enrollment: 3859 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Locations of femoral fracture | up tp 2 months
  To provide a summary of covariate information regarding the occurrence of femur Fractures at a specific site.

CONTACTS AND LOCATIONS:
Overall Officials: TSANG-TANG Hsieh, MD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan